CLINICAL TRIAL: NCT03012568
Title: ASSURE MRI Study - Clinical Study to Confirm MRI Safety and Effectiveness Using St. Jude Medical (SJM) Cardiac Rhythm Management Systems
Brief Title: Clinical Study to Confirm MRI Safety and Effectiveness Using St. Jude Medical (SJM) Cardiac Rhythm Management Systems
Acronym: ASSUREMRI
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10137
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Bradycardia; Tachycardia
MeSH Terms: conditions — Bradycardia; Tachycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SJM Implantable cardiac devices — SJM implantable devices undergoing MRI scan
  Other Names: ICD; CRT-D; Pacemakers; CRT; MRI; Leads

SUMMARY:
This is a clinical investigational plan (CIP) for the "Clinical Study to Confirm MRI Safety and Effectiveness Using SJM Cardiac Rhythm Management Systems (ASSURE MRI)". This study intends to enroll patients who meet standard bradycardia or tachycardia indications and have already been implanted with one of the SJM device/lead combinations listed in this protocol. The objective of this study is to confirm the safety and effectiveness of each of the four SJM device/lead combinations in an MRI environment. This clinical investigation is sponsored by St. Jude Medical.

DETAILED DESCRIPTION:
This is a prospective, multi-center clinical study designed to confirm the safety and effectiveness of St. Jude Medical low voltage pacemakers, high voltage dual chamber Implantable Cardioverter-Defibrillators (ICD), and Cardiac Resynchronization Therapy Defibrillators (CRT-D) with various leads in an MRI environment.

The study will enroll subjects across multiple geographies and sites. Sites in geographies where MRI labelling is not yet approved may also be included after appropriate IRB/EC and local regulatory approvals, as applicable, are obtained. A prospective, multi-center study design is chosen for generalizability of study results.

The clinical study will be conducted in approximately 40 centers worldwide. Approximately 88 subjects total (with a minimum 22 subjects for each of the four device/lead combinations) will be enrolled in this study.

Enrollment in the study is expected to take approximately 6-8 months. Subjects will be followed for 1 month following the MRI scan. The total study duration of the study is expected to be 10 months, depending on the rate of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Are implanted with one of the following SJM device/lead combinations evaluated in this study for at least 60 days (can include patients with an eligible SJM lead for ≥ 60 days OR patients with a new eligible SJM pacemaker, Implantable Cardioverter-Defibrillators (ICD), or Cardiac Resynchronization Therapy Defibrillators (CRT-D) device and eligible SJM lead implanted for at least 60 days:

  1. Accent MRI™, Assurity MRI™, Endurity MRI™, or Endurity pacemaker with Tendril™ STS Model 2088 lead
  2. Accent MRI™, Assurity MRI™, Endurity MRI™, or Endurity pacemaker with IsoFlex™ Optim (Model 1944 or 1948) lead
  3. Ellipse™ VR/DR or Fortify Assura VR/DR ICD with Tendril™ STS (Model 2088) or Tendril MRI™ and Durata™ or Optisure™ leads
  4. Quadra Assura™ CRT-D with Tendril™ STS (Model 2088), Durata™ or Optisure™, and Quartet™ Quadripolar leads
* Are implanted with an eligible SJM pacemaker, ICD, or CRT-D device pectorally
* Be willing to undergo an elective MRI scan without sedation. Note: Antianxiety agents (e.g. minor tranquilizers, etc.) may be used as long as the subject can communicate with site personnel during the MRI scan
* Be able to provide informed consent for study participation (legal guardian is NOT acceptable)
* Be willing and able to comply with the prescribed follow-up tests and schedule of evaluations

Exclusion Criteria:

* Have another existing active implanted medical device, e.g., neurostimulator, infusion pump, etc. that has MR labeling that will not allow the MRI scans per this protocol to be completed.
* Have other non-MRI compatible device or material implanted

  * NOTE: MRI compatible knee replacements, hip replacements, stents, etc. may be included as long as the labeling of these devices allow MRI scans conducted per this protocol
  * NOTE: MRI compatible mechanical, prosthetic, and bioprosthetic heart valves may be included as long as the labeling of these devices allow for MRI scans conducted per this protocol
  * NOTE: Non-removable dental implants may be included
* Have a lead extender, adaptor, or capped/abandoned lead
* Be unable to fit in MRI bore, i.e., subject will come into contact with the magnet façade inside the MRI bore.
* Are currently participating in a clinical investigation that includes an active treatment arm
* Are pregnant or planning to become pregnant during the duration of the study
* Have a life expectancy of less than 3 months due to any condition
* Meet exclusion criteria per local law (e.g. age)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who meet standard bradycardia or tachycardia indications comprise the target population for this study. The subject will be considered enrolled in the study after the consent is signed and the MRI Settings have been programmed at the MRI visit.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint: Freedom from MRI scan-related complications | One month following the MRI scan.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Kim, Study Director — Abbott Medical Devices
Locations (3):
- Australia (2):
  - Heart Care Partners - Wesley Hospital, Auchenflower, Queensland
  - Heart Care Western Australia, Perth, Western Australia
- CARE Banjara, Hyderabad, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided